CLINICAL TRIAL: NCT04862897
Title: Patient-controlled Admissions to Inpatient Care for Patients With Severe Psychiatric Conditions in Region Stockholm
Brief Title: Patient-controlled Admissions to Inpatient Care
Status: Recruiting | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: Stockholm Health Care Services (Unknown)
Responsible Party: Principal Investigator, Alexander Rozental, Principal investigator, Karolinska Institutet
Other Study IDs: 2020-06498
Record Dates: First submitted 2021-04-20; First posted 2021-04-28 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Patient-controlled Admissions; Matched Control Group
Keywords: Patient-controlled admissions; Self-referrals; Patient participation; Inpatient care
MeSH Terms: conditions — Patient Participation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patient-controlled admissions: Patients who have been granted access to patient-controlled admissions
  Interventions: Other: Patient-controlled admissions
- Matched control group: Patients matched on account of age, gender, diagnosis, and history of psychiatric inpatient care, but who have not been granted access to patient-controlled admissions

INTERVENTIONS:
Other: Patient-controlled admissions — Patients are allowed to admit themselves to inpatient care when needed (standard procedure, four days of inpatient care at a time, up to three times a month)
  Groups: Patient-controlled admissions

SUMMARY:
Patient-controlled admissions refer to the possibility for patients with severe psychiatric conditions to admit themselves to inpatient care. Compared to having the healthcare providers make this decision, patient-controlled admissions are believed to decrease the need for involuntary care, decrease symptom levels, and increase quality of life and autonomy for the patient. The current research project aims to evaluate the implementation of patient-controlled admissions to all patients with severe psychiatric conditions within Region Stockholm, Sweden, including child and adolescent psychiatry (but excluding forensic psychiatry and addiction care).

DETAILED DESCRIPTION:
Patients with severe psychiatric conditions represent a group who have extensive care needs and for whom few effective interventions exist. Diagnoses such as schizophrenia and borderline personality disorder usually have a poor prognostic outlook in terms of recovery, and patients often suffer from life-long disabilities. Meanwhile, their healthcare expenditures are typically high. In case of increased symptoms and novel sickness spells, healthcare providers make an assessment if admission to inpatient care is needed. This gatekeeper-model is typical of most western countries and infers that the decision to be admitted is always made by a third party. Since about a decade, attempts at transferring the responsibility of admissions to patients themselves is being implemented and tested in several countries and contexts, referred to as patient-controlled admissions. The idea is to increase patient involvement, enhance self-determination, and improve their ability to manage signs of illness. Patient-controlled admissions involve signing an agreement between inpatient care, outpatient care, and those patients that are deemed to have the highest care needs, whereby the patients can contact an inpatient ward and be admitted when required. Previous research has revealed that patient-controlled admissions decrease involuntary admissions and that both healthcare providers and patients are positive towards its use. These studies have however been small and used limited outcome measures. The current research project aims to study the results of implementing patient-controlled admissions to all patients with severe psychiatric conditions within Region Stockholm, Sweden, including child and adolescent psychiatry (but excluding forensic psychiatry and addiction care). Apart from determining the possible impact on both number of admissions and days in admission (voluntary and involuntary), other psychiatric or somatic healthcare consumption, sick-leave, and redeemed medical prescriptions, self-report measures will be used to assess the effects on symptom levels, quality of life, and autonomy. A matched control group (matched on account of age, gender, diagnosis, and history of psychiatric inpatient care, but who have not been granted access to patient-controlled admissions) will also be utilised to determine the effects of patient-controlled admissions on all primary outcomes measures, other psychiatric or somatic healthcare consumption, sick-leave, and redeemed medical prescriptions.

ELIGIBILITY:
Inclusion Criteria:

* Have an on-going contact with outpatient care.
* Have an individual care plan and crisis plan.
* Have had at least one inpatient care period the previous year.
* Are expected to have the greatest need of inpatient care.
* Are interested in, and understand the concept of, patient-controlled admissions.

Exclusion Criteria:

* No informed consent to participate in the research project (concerns only self-reported outcomes).

Matched control group:

- A matched control group consisting of seven times the number of of patients receiving patient-control admissions will be utilised for all primary outcome measures, other psychiatric or somatic healthcare consumption, sick-leave, and redeemed prescriptions (matched on account of age, gender, diagnosis, and history of psychiatric inpatient care, but who have not been granted access to patient-controlled admissions)

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with severe psychiatric conditions in Region Stockholm who fulfil the inclusion criteria can be provided access to patient-controlled admissions. This includes child and adolescent psychiatry, but excludes forensic psychiatry and addiction care. All patients who receives patient-controlled admissions and a matched control group will be evaluated regarding all primary outcome measures, other psychiatric or somatic healthcare consumption, sick-leave, and redeemed medical prescriptions. For the remaining secondary outcomes measures (i.e., self-reported outcomes), only those patients who consent to participate in the research project will be evaluated.
Sampling Method: Non-Probability Sample
Enrollment: 564 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Admissions to inpatient care | Change in number of admissions to inpatient care between baseline and at 12 months
  Number of admissions to inpatient care
Days in inpatient care | Change in number of days in inpatient care between baseline and 12 months
  Number of days in inpatient care
Admissions to inpatient care | Change in number of admissions to inpatient care between baseline and at 24 months
  Number of admissions to inpatient care
Days in inpatient care | Change in number of days in inpatient care between baseline and 24 months
  Number of days in inpatient care
Admissions to inpatient care | Change in number of admissions to inpatient care between baseline and at 36 months
  Number of admissions to inpatient care
Days in inpatient care | Change in number of days in inpatient care between baseline and 36 months
  Number of days in inpatient care
Admissions to involuntary care | Change in number of admissions to involuntary care between baseline and at 12 months
  Number of admissions to involuntary care
Days in involuntary care | Change in number of days in involuntary care between baseline and at 12 months
  Number of days in involuntary care
Admissions to involuntary care | Change in number of admissions to involuntary care between baseline and at 24 months
  Number of admissions to involuntary care
Days in involuntary care | Change in number of days in involuntary care between baseline and at 24 months
  Number of days in involuntary care
Admissions to involuntary care | Change in number of admissions to involuntary care between baseline and at 36 months
  Number of admissions to involuntary care
Days in involuntary care | Change in number of days in involuntary care between baseline and at 36 months
  Number of days in involuntary care
Coercive measures | Change in number of coercive measures between baseline and at 12 months
  Number of coercive measures (forced medication, seclusion, and restraint)
Coercive measures | Change in number of coercive measures between baseline and at 24 months
  Number of coercive measures (forced medication, seclusion, and restraint)
Coercive measures | Change in number of coercive measures between baseline and at 36 months
  Number of coercive measures (forced medication, seclusion, and restraint)

SECONDARY OUTCOMES:
EQ5D-5L | Change in self-rated quality of life (somatic) between baseline and at 12 months
  Self-rated quality of life (somatic) on five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has five levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The scores for the five dimensions can be combined into a five-digit number that describes the patient's health state, with 11,111 indicating perfect health and 55,555 the worst health state. The outcome ranges from 5 (no health limitations at all, 11,111) to 25 (for state 55,555).
World Health Organization Disability Assessment Schedule | Change in self-rated quality of life (somatic) between baseline and at 12 months
  Self-rated quality of life (somatic) on six dimensions: cognition, mobility, self-care, getting along with people, life activities and participation - including work-related disability. The scores assigned to each of the items - "none" (1), "mild" (2) "moderate" (3), "severe" (4) and "extreme" (5) - are then summed. A higher sum score indicates worse quality of life (100 = full disability; 0 = no disability).
Clinical Global Impression | Change in clinician-rated functional level between baseline and at 12 months
  Clinician-rated functional level, measuring symptom severity, treatment response and the efficacy of treatments in treatment studies of patients with mental disorders. It has two domains, severity scale and Improvement scale. Both are scored on a 7 point scale; 1 = Normal, not at all ill to 7 = Among the most extremely ill patients, as well as 1 = Very much improved, and 7 = Very much worse. A higher score indicates worse functional level and a worsening of functioning, respectively.
Brunnsviken Brief Quality of life scale | Change in self-rated quality of life (psychological) between baseline and at 12 months
  Self-rated quality of life (psychological), including 12 items covering six life areas: Leisure, View on life, Creativity, Learning, Friends and Friendship, and View on self. All items are scored using the same response format, con- sisting of a five-step Likert rating scale, visually scored 0-4 with written anchor points at 0 (Strongly disagree) and 4 (Strongly agree). The BBQ total score is computed by summing the weighted satisfaction ratings, i.e. by multiplying the Satisfaction and Importance items for each life area and summing the six products for a total score (possible score range 0-96). A higher sum score indicates a better quality of life.
General Self-Efficacy scale | Change in self-rated self-efficacy between baseline and at 12 months
  Self-rated self-efficacy, assessing a general sense of perceived self-efficacy with the aim in mind to predict coping with daily hassles as well as adaptation after experiencing all kinds of stressful life events. The response to 10 items are made on a 4-point scale ( 1 = Not at all true, 2 = Hardly true, 3 = Moderately true. 4 = Exactly true). The sum of all 10 items yield the final composite score with a range from 10 to 40. A higher sum score indicates a higher self-efficacy.
Generalized Anxiety Disorder - 7 items | Change in self-rated anxiety between baseline and at 12 months
  Self-rated anxiety, a seven-item instrument that is used to measure or assess the severity of generalised anxiety disorder and symptoms of anxiety and worry. The GAD-7 score is calculated by assigning scores of 0, 1, 2, and 3, to the response categories of "not at all," "several days," "more than half the days," and "nearly every day," respectively, and then adding together the scores for the seven questions. GAD-7 total score for the seven items ranges from 0 to 21. Scores of 5, 10, and 15 represent cut-points for mild, moderate, and severe anxiety, respectively.
The Patient Health Questionnaire - 9 items | Change in self-rated depression between baseline and at 12 months
  Self-rated depression, measures depression using nine items on 4-point scales and a 4-point scale for impact on daily life. As a severity measure, the PHQ-9 score can range from 0 to 27, since each of the 9 items can be scored from 0 (not at all) to 3 (nearly every day); 0-4 = minimal depression, 5-9 = mild depression, 10-14 = moderate depression, 15-19 = moderately severe depression, 20-27 = severe depression.
Visual Analogue Scales | Change in self-rated care needs and current health status between baseline and at 12 months
  Four items assessing different aspects of the patients' care needs and current health status are administered monthly. These include the following; 1) "I feel confident about receiving care when I need it" 2) "I am able to actively participate in my care", and 3) "I believe care is available when needed". These are scored on a continuum ranging from "I do not agree at all" (0) to "Totally agree" (10). Also, a fourth item concerns "How would you rate your current health status?", which is rated between "Worst possible health" (0) and "Best possible health" (10).
Other psychiatric or somatic healthcare consumption | Change in number of other psychiatric or somatic healthcare consumption between baseline and 12 months
  Number of other psychiatric or somatic healthcare consumption
Sick-leave | Change in number of days in sick-leave between baseline and 12 months
  Number of days in sick-leave
Redeemed medical prescriptions | Change in number of redeemed medical prescriptions between baseline and 12 months
  Number of redeemed medical prescriptions

OTHER OUTCOMES:
KIDSCREEN | Change in self-rated quality of life (health-related) between baseline and at 12 months
  For child and adolescent psychiatry only: Self-rated quality of life (health-related), using 11 items. It is scored on a five-point Likert-scale, "Not at all" or "Never" (0) to "Extreme" or "Always" (4). One item is supposed to reflect the participant's overall health status, i.e., "In general, how would you say your health is?". KIDSCREEN is administered to both the patients and their caregivers.
Alcohol, Smoking and Substance Involvement Screening Test | Change in self-rated alcohol and substance use between baseline and at 12 months
  For child and adolescent psychiatry only: Self-rated alcohol and substance use, using 7 items. Item 1 has a no/yes-response, items 2-5 has a 0, 5, 6, 7, 8 scale, ranging from "Never" to "Daily or almost daily", item 6 has a 0, 6, 3 scale, ranging from "No, never" to "Yes, but not in the past 3 months", and item 7 has a categorical respons "No, never", "Yes, the past 3 months", and "Yes, but not in the past 3 months". Scores from items 2-6 are summed, with a higher score indicating greater severity of alcohol, smoking, and substance use.
Childrens Global Assessment Scale | Change in clinician-rated functional level between baseline and at 12 months
  For child and adolescent psychiatry only: Clinician-rated functional level. The child or young person is given a single score between 1 and 100, based on a clinician's assessment of a range of aspects related to a child's psychological and social functioning. The score will put them in one of ten categories that range from 'extremely impaired' (1-10) to 'doing very well' (91-100): 0-10: Extremely impaired (24 hour care), 11-20: Very severely impaired, 21-30: Severe problems, 31-40: Serious problems, 41-50: Obvious problems, 51-60: Some noticeable problems, 61-70: Some problems, 71-80: Doing all right, 81-90: Doing well, 91-100: Doing very well.
The Strengths and Difficulties Questionnaire | Change in self-rated functional level between baseline and at 12 months
  For child and adolescent psychiatry only: Self-rated functional level that ask about 25 attributes, some positive and others negative. These 25 items are divided between 5 scales: emotional symptoms (5 items), conduct problems (5 items), hyperactivity/inattention (5 items), peer relationship problems (5 items), prosocial behaviour (5 items). The four first scales generate a totalt difficulties score, with a higher score indicating greater difficulties (0-40). The Strengths and Difficulties Questionnaire is administered to both the patients and their caregivers.
Revised Children's Anxiety and Depression Scale | Change in self-rated anxiety and depression between baseline and at 12 months
  For child and adolescent psychiatry only: Self-rated anxiety and depression, a 47-item, youth self-report questionnaire with subscales including: separation anxiety disorder, social phobia, generalized anxiety disorder, panic disorder, obsessive compulsive disorder, and low mood (major depressive disorder). It also yields a Total Anxiety Scale (sum of the 5 anxiety subscales) and a Total Internalizing Scale (sum of all 6 subscales). A higher score indicates greater symptom severity. The Revised Children's Anxiety and Depression Scale is administered to both the patients and their caregivers.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Rozental, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Centre for Psychiatry Research, Stockholm, Stockholm County, Sweden

IPD SHARING:
Plan to Share IPD: No
Data include patient records and need a permit from Stockholm Health Care Services in order to become available to other researchers.

REFERENCES:
- [Background] Smitmanis Lyle M, Allenius E, Salomonsson S, Bjorkdahl A, Strand M, Flyckt L, Hellner C, Lundgren T, Jayaram-Lindstrom N, Rozental A. What are the effects of implementing patient-controlled admissions in inpatient care? A study protocol of a large-scale implementation and naturalistic evaluation for adult and adolescent patients with severe psychiatric conditions throughout Region Stockholm. BMJ Open. 2022 Aug 16;12(8):e065770. doi: 10.1136/bmjopen-2022-065770. PMID 35973700
- See also: Related Info — https://www.psykiatriforskning.se/utveckling/verksamhetsutveckling-psykiatri/sjalvvald-inlaggning/